CLINICAL TRIAL: NCT05567302
Title: Immediate Effect of Cervical Manual Therapy Methods in Patients With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cervical Manual Therapy
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Neck Pain
Keywords: manuel therapy; neck
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations; Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Evaluation and treatment will be carried out by different physiotherapists. In this way, it is aimed to provide an objective evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy (Experimental): Manual therapy, manipulative therapy, is a completely manual treatment method that includes special techniques and is known as a treatment that aims to correct bony deformities and is highly effective when combined with exercise.
  Interventions: Other: Manual therapy
- myofascial release (Active Comparator): Foam rollers are a popular tool for helping athletes release muscle knots or trigger points.Myofascial release is a soft tissue method that provides removal of adhesions and tissue tension in tissues due to overload and repetitive use.
  Interventions: Other: myofascial release

INTERVENTIONS:
Other: Manual therapy — In lower cervical lateral flexion problems, manipulative correction technique will be applied from the articular pillar part of the superior vertebra on the side where the limitation is present.
  In lower cervical lateral flexion problems, manipulative correction technique will be applied from the articular pillar part of the superior vertebra on the side where the limitation is present.
  A rotational maneuver will be performed from the posterior side of the articular pillar part of the superior vertebra, on the opposite side of the side where the movement restriction is present.
  Arms: Manual therapy
Other: myofascial release — The soft tissue is palpated by the physiotherapist and pressure is applied directly to the skin until the tissue barrier is felt in the direction of restriction. Once the tissue barrier is present, it is applied for 90-120 seconds, without slipping on the skin or forcing the tissue, until the fascia complex begins to loosen and a softening sensation is achieved.
  Arms: myofascial release

SUMMARY:
Chronic neck pain is an important health problem in modern society and is frequently encountered today. Approximately 10% of the adult population experiences neck pain at least once in their lives.

Anamnesis of the patient with neck pain; It should include the patient's complaints, illness history, family history, social status, work life and leisure activities.

The age of the patient, the severity of the symptoms, the mechanism of the injury, the activity history, the duration of the symptoms, the location and limits, the spread of the pain, the relationship of the complaints with the change in position, the restrictions during movement, and the sleeping positions should be taken into account. In addition, past diseases, operations and current diseases, medications used should be recorded.

Among chronic pains, neck pain ranks second after low back pain. Physical stresses in daily living activities, maintaining static posture and sleeping habits, carrying bags and weights in the wrong position, muscle imbalance are important factors in neck pain. Although cervical spine involvements have a great effect on neck pain, almost all of them have paravertebral muscle spasm, especially trapezius muscle spasm. Physiotherapy applications are widely used in the treatment of chronic neck pain.

DETAILED DESCRIPTION:
Therapeutic approaches are frequently used to reduce inflammation and accelerate the healing process. Reducing pain in neck diseases, ensuring sufficient length of the muscle, strength balance, improving strength and function, improving postural re-education and cervical movements are the main goals. With the increasing prevalence of neck pain, the search for new treatment methods is increasing.

It includes manual therapy, manipulation, acupuncture, and soft tissue therapy for chronic neck pain. Neck pain results from deep muscle dysfunctions and altered fascia structures. In this case, it may cause the disruption of the continuous musculofacial corset-like system. In addition, changes in the fascia (increased fascial thickness and disruption of fascial alignment) may affect this system more. Myofascial release is one of the soft tissue treatment applications. Although there are studies reporting that myofascial release is a method that can achieve positive effects such as reducing pain intensity and improving muscle function, there are few studies on this subject in the literature and sufficient evidence has not been reached.

ELIGIBILITY:
Inclusion Criteria:

* Neck pain
* Being between 20-60 years old

Exclusion Criteria:

* Cardiopulmonary disease
* malignancy and pregnancy
* Operation, injection, etc. for the neck in the last 3 months. those with a history of treatment
* Spine surgery
* Psychological discomfort
* Neurological and orthopedic deficits

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2022-10-08 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | one day
  In the measurement of neck pain severity, a standard, proven reliability 10 mm VAS will be used. A value between 0 and 10 will be determined for the VAS, with 0 in the absence of pain and 10 mm in the most severe pain.
pinchmeter | one day
  Finger grip strength is evaluated with a pinchmeter in both hands. Prior to measurements, participants will be verbally informed and allowed to experiment. When the participants are ready, they are asked to squeeze the dynamometer with all their strength for 3 seconds and then release it. Participants will rest for 1 minute between measurements. The same process is repeated in the same way after the application and the values are noted.
Jamar Hand Dynomometer | one day
  The grip strengths of all participants were in the standard position recommended by the "American Society of Hand Therapist" on both hands; Hand dynamometer is evaluated with elbow in 90° flexion, forearm and wrist in neutral position. When participants are ready, they will be asked to squeeze the dynamometer with all their strength for 3 seconds and then release it. Rest for 1 minute between measurements. The evaluation will be taken three times and the averages will be recorded as a result of the measurement. The same process is repeated in the same way after the application and the values are noted.

SECONDARY OUTCOMES:
Scoliometer | one day
  Bending the patient forward about 45 degrees is the angle at which the rotational deformity in the back region is best seen. The evaluation is completed by reading the degree of rotation of the curvature on the scoliometer according to the level where the curvature is highest.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol hospital, Istanbul, Istanbul Avrupa Kitasi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghan GM, Babu VS. Immediate Effect of Cervico-thoracic Mobilization on Deep Neck Flexors Strength in Individuals with Forward Head Posture: A Randomized Controlled Trial. J Man Manip Ther. 2021 Jun;29(3):147-157. doi: 10.1080/10669817.2020.1834321. Epub 2020 Oct 22. PMID 33090945